CLINICAL TRIAL: NCT05607134
Title: Effect of Radial Extracorporeal Shock Wave and Peripheral Magnetic Stimulation on Upper Limb in Children With Spastic Hemiplegia
Brief Title: Effect of Extracorporeal Shock Wave and Peripheral Magnetic Stimulation on Spastic CP Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Abdelaziz Saad, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 012/003862
Record Dates: First submitted 2022-10-27; First posted 2022-11-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Hemiplegic Cerebral palsy; Radial Extracorporeal Shock Wave; Peripheral magnetic stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical and occupational therapy group (Sham Comparator): The group will receive a Physical and occupational therapy program
  Interventions: Other: selected physical and occupational therapy program
- Shock Wave group (Active Comparator): The group will receive a radial Extracorporeal Shock Wave sessions
  Interventions: Device: Radial Extracorporeal Shock Wave
- Peripheral Magnetic Stimulation group (Active Comparator): The group will receive a Peripheral Magnetic Stimulation sessions
  Interventions: Device: Peripheral magnetic stimulation

INTERVENTIONS:
Other: selected physical and occupational therapy program — The children in this group will receive a selected physical and occupational therapy programs one hour three times weekly for eight successive weeks.
  Arms: Physical and occupational therapy group
Device: Radial Extracorporeal Shock Wave — The children in this group will receive in addition to the selected physical therapy and occupational program as single session of shock wave intervention once per week for four eight successive weeks using (STORZ MEDICAL AG, Tagerwilen, Schweiz) device. rESWT will be applied on flexor carpi ulnaris, flexor carpi radialis, in the middle of the muscle belly and tendons of flexor digitorum on the palm. The treatment protocol of rESW will follow; 1500 shoots for each muscle; 0.030 mj/mm2; 4 HZ with pressure 1 bar will be used.
  Arms: Shock Wave group
Device: Peripheral magnetic stimulation — The children in this group will receive in addition to the selected physical therapy program peripheral magnetic stimulation (PMS) therapy for twenty minutes, three sessions per week, for eight successive weeks using Peripheral magnetic stimulation device "A MAGNUM XL Pro, Globus, Italia". The PMS consisted of 2000 stimuli at a stimulation frequency of 20Hz, a train duration of 1 second, and an intertrain interval of 2 seconds. Intensity was individually set at 10% to 100% of the maximum stimulus intensity.
  Arms: Peripheral Magnetic Stimulation group

SUMMARY:
Hypotheses:

There will be an effect of radial extracorporeal shock wave therapy and peripheral magnetic stimulation on the following parameters, in children with spastic hemiplegia:

* Wrist flexors spasticity.
* Wrist joint range of motion.
* Hand grip muscles strength.
* Sensorimotor function of wrist and hand.

DETAILED DESCRIPTION:
Significance of the study:

Reducing muscle hypertonia or spasticity in order to regain independent mobility is an essential goal of a physiotherapeutical treatment in neuro-rehabilitation. The rapid normalization of the muscle tone is a criterion that can crucially influence the outcome of future rehabilitation or in training programs.

Purposes of the study:

To evaluate the effect of radial extracorporeal shock wave therapy and peripheral magnetic stimulation on the following parameters, in Children with Spastic Hemiplegia:

* Wrist flexors spasticity.
* Wrist joint range of motion.
* Hand grip muscles strength.
* Sensorimotor function of wrist and hand.

Methods:

Forty-five children with hemiplegic cerebral palsy, aged from 6 to 10 years, will be enrolled in this study. Wrist flexors spasticity, Wrist joint range of motion, Hand grip muscles strength, Sensorimotor function of wrist and hand will be assessed.

Data Analysis and statistical design:

Normally distributed numerical data will be statistically described in terms of mean standard deviation, while not-normal data will be represented as median and range or inter-quartile range (IQR). Qualitative (categorical) data will be described in frequencies (number of cases) and percentage. Numerical data will be tested for the normal assumption using Kolmogorov Smirnov test.

Comparison of numerical variables between the study groups will be done using One Way Analysis of variance (ANOVA) test when normally distributed and Kruskal Wallis analysis of variance (ANOVA) test when not normal.

For comparing categorical data, Chi-square test will be performed. Exact test will be used instead when the expected frequency is less than 5.

A probability value (p value) less than 0.05 is considered statistically significant. All statistical calculations will be done using computer programs Microsoft Excel 2019 (Microsoft Corporation, NY, USA) and IBM SPSS (Statistical Package for the Social Science; IBM Corp, Armonk, NY, USA) release 22 for Microsoft Windows.

ELIGIBILITY:
Inclusion Criteria:

* • Spastic hemiplegic children will be included in this study.

  * The children ages will be ranged from 6-10 years chronologically.
  * Children will have wrist flexors degree of spasticity ranged from +1 to 2 on Modified Ashworth Scale.
  * The children will have Level III to Level IV according to the Manual Ability Classiﬁcation System.
  * All children will be medically stable.
  * Children take their anti-spasticity medications.
  * All children will be able to follow instructions.

Exclusion Criteria:

* • History of recent nonunion fracture of the upper extremities.

  * Neurological or orthopedic surgery in the upper extremities in the last 12 months before the study.
  * Received Botulinum toxin A injections in the last six months.
  * Fixed contractures and deformities.
  * Patients with a self-contained medical implant such as: a metal plate along the spastic limbs, pacemaker, cochlear implant, and so on.
  * Children with cognitive dysfunction.
  * Poor skin integrity.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change of the muscle tone of the wrist flexors | at the beginning and after eight weeks of the intervention
  The muscle tone of the wrist flexors will be assessed with The Modified Tardieu Scale (MTS) . This test is done in the supine position, with head in midline, and is measured at 3 different velocities (V1, V2, and V3). V1: as slow as possible (slower than the natural drop of the limb segment under gravity. V2: speed of limb segment falling under gravity. V3: as fast as possible faster than the rate of the natural drop of the limb segment under gravity. Measuring R1 (the fast velocity movement of the wrist through the full ROM to determine the point of catch in the ROM), R2 (the passive ROM), and R2-R1 (dynamic component of spasticity).

SECONDARY OUTCOMES:
Change of wrist extension range of motion (ROM) | at the beginning and after eight weeks of the intervention.
  Wrist extension will be measured for all children according to Norkin and White (2016) as follows: Each child was placed in sitting next to a supporting surface with the elbow flexed to 90 degrees, and the palm of the hand facing the ground. The forearm was rested on the supporting surface, but the hand was leaved free to move without radial or ulnar deviation of the wrist. The children were asked to extend the wrist by moving the hand in a dorsal direction toward the ceiling with maintaining the wrist in 0 degrees of radial and ulnar deviation.
  Goniometer alignment:
  1. Fulcrum of the goniometer was placed on the lateral aspect of the wrist over the triquetrum.
  2. Proximal arm was aligned with the lateral midline of the ulna, using the olecranon and ulnar styloid process for reference.
  3. Distal arm was aligned with the lateral midline of the fifth metacarpal.
Change of handgrip strength | at the beginning and after eight weeks of the intervention.
  The isometric muscle strength of hand grip will be measured with a handheld dynamometer. The position of the dynamometer will be standardized for each measurement. A 'make' test will be employed with the tester setting a constant resistive force for 3 to 5 seconds, directed perpendicular to the long axis of the limb segment to elicit an isometric muscle contraction. A standard instruction of 'close your hand as hard as you can' is given to each participant for each trial (Berry et al., 2004).
  Children will be given two practical trials until the investigator will be confident that they understand the task. Each child will perform three trials, strong verbal encouragement will be used during the trial to achieve maximum effort and the peak force values from dynamometer will be recorded (Thompson et al., 2011).
Change of Functionality of wrist and hand | at the beginning and after eight weeks of the intervention.
  The upper extremity section of the Fugl-Meyer Assessment (FMA-UE) is used. The FMA-UE wrist and hand motor and sensory subscores are graded, and the scores are added (total 36 scores). Each domain contains multiple items, each scored on a 3-point ordinal scale (0, cannot perform; 1, performs partially; 2, performs fully) (Fugl-Meyer et al., 1975; Krewer et al., 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Hany A. Saad, M. SC., Principal Investigator — Cairo University; KHALED A. MAMDOUH, PHD, Study Chair — Prof. of Physical Therapy for Pediatrics, Faculty of Physical Therapy, Cairo University; Hoda A. EL-TALAWY, PHD, Study Director — Prof. of Ph.Th. for Pediatrics, Faculty of Physical Therapy, Cairo University; Mohamed A. Elshafey, PHD, Study Director — Ass. Prof. of Physical Therapy for Pediatrics, Faculty of Physical Therapy, Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt